CLINICAL TRIAL: NCT03183505
Title: Safety and Efficacy Study of Anyu Peibo in the Treatment of Major Depressive Disorder(MDD): a Ⅱb Stratified Randomized, Double-Blind, Placebo-Paralleled, Multicenter Clinical Trial
Brief Title: Comparison of Anyu Peibo With Placebo in Treatment of MDD，Ⅱb
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Su Zhou YiHua Biotechnology Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYPB-MDD-Ⅱb-1701; 2017ZX09304-020 (Other Grant/Funding Number: China National Major Project for IND)
Record Dates: First submitted 2017-06-05; First posted 2017-06-12 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anyu Peibo (Experimental): Anyu Peibo Capsule, oral, 0.8g twice per day
  Interventions: Drug: Anyu Peibo
- Placebo (Placebo Comparator): Placebo,oral, twice per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anyu Peibo — Anyu Peibo Capsule, 0.8g twice per day, oral after breakfast and supper
  Other Names: Anyu Peibo Capsule
  Arms: Anyu Peibo
Drug: Placebo — Placebo Capsule, twice per day, oral after breakfast and supper
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Anyu Peibo Capsule comparing with placebo in the treatment of Chinese Patients with Depression. And to provide some scientific evidence for protocol designing in following phase Ⅲ clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult with primary diagnosis of major depressive disorder(MDD) based on the criteria of DSM-5, single episode or recurrent episode.
* The total score of MADRS is ≥24 in both screening visit and baseline visit.
* The total score of HAMD-17 is ≥18 and the first item (depressed mood) is ≥2 in both screening visit and baseline visit.
* CGI-S is ≥4 in both screening visit and baseline visit.
* The subject understands and consents to takes part in this clinical trials. The subjects should sign informed consent form.

Exclusion Criteria:

* The subject has a suicide attempt within recent 1 year, or has a currently significant risk of suicide, or has a score ≥3 on item 3(suicide assessment) of the HAMD.
* The subject has a current psychiatric diagnosis other than depression.
* When the HAMD-17 score of baseline visit compares with the screening visit, the decreasing rate is ≥25%.
* Known hypersensitivity to Big Leaf Ju, or at least to two kinds of drugs.
* Any unstable cardiovascular, hepatic, renal, blood, endocrine, or other medical disease.
* Any neurological disease (such as Parkinson's Disease, cerebrovascular accident and epilepsy) or cerebral injury (traumatic or disease related).
* Had a history or a high risk related disease or medication of seizure disorder,except infantile febrile convulsion.
* Had a history of hyperthyroidism or hypothyroidism within recent 1 year and still taking medication.
* With psychotic symptoms.
* The subject has a history of mania episode, including manic, mixed, bipolar depression or rapid cycle attack.
* The subject has a current diagnosis of depression due to a somatic disease.
* The subject could not take medication or has a disease affecting drug absorption, such as active bowel disease, partial or total intestinal obstruction, or chronic diarrhea.
* Clinically significant electrocardiographic(ECG) abnormalities in screening visit. Such as QTc ≥450 ms in male or ≥470 ms in female; Sinus bradycardia and HR ≤ 50 bpm; Ⅲ atrioventricular block; atrial fibrillation, etc.
* Clinically significant abnormal laboratory values(eg. Routine blood value above or below 1.2 times of the normal range; urine WBC, RBC or protein ≥++; ALT or AST value above 1.5 times of clinical top-limit; BUN value above 1.2 times of top-limit; Cr value above normal top-limit; thyroid gland function index above or below 1.2 times of the normal range, Fasting plasma glucose value above 1.2 times of normal top-limit; blood fat value above 1.5 times of normal top-limit).
* The subject who used at least two different antidepressants with recommended dose and adequate duration (maximum dosage by at least 4 weeks according to label) treatment still had no respond.
* The subject uses antidepressant drug normally before 2 weeks of screening, and stops using psychotropic drug before randomization less than 7 half-life period (monoamine oxidase inhibitor: at least 2 weeks; fluoxetine: at least 1 month)
* The subject received light therapy within 2 weeks.
* The subject received ECT, trans-cranial magnetic stimulation, or other physics therapy within 3 months.
* The subject received systematic psychotherapy (interpersonal relationship, psychoanalytic therapy, or cognitive behavioral therapy) within 3 months or plan to use systematic psychotherapy during the study period.
* The subject has a history of substance abuse (including alcohol, drug or other psychoactive substance) within 1 year before screening.
* Women who were pregnant, breast-feeding, or serum-HCG(+) on screening; or planning to become pregnant within 3 months after kick-off of clinical trial.
* The subject has participated in a drug clinical trial within 1 month before screening.
* The investigator thinks the subject is unsuitable to enroll in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
The change of total score from baseline in MADRS scale | 6 weeks

SECONDARY OUTCOMES:
Clinical Response Rate according to MADRS | 6 weeks
Clinical Remission Rate according to MADRS | 6 weeks
Clinical Response Rate according to HAMD-17 | 6 weeks
Clinical Remission Rate according to HAMD-17 | 6 weeks
the Change of CGI (CGI-S, CGI-I) from baseline | 6 weeks
the Change of total score from baseline in HAMA | 6 weeks
  Hamilton Anxiety Rating Scale

OTHER OUTCOMES:
Physical Examination | 6 weeks
AE | 6 weeks
  Adverse Events
Laboratory Examination | 6 weeks
  Blood RT, Urinalysis, Hepatic function, Renal function, FBG, Lipid, CK, Thyroid Function Test and Serum-HCG(fertile women only)
the Change of ECG from baseline | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (8):
- China (8):
  - Beijing Anding Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Jiangxi Mental Hospital, Nanchang, Jiangxi
  - Brain Hospital of Jilin Province, Siping, Jilin
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - XI'AN Mental Health Center, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan